CLINICAL TRIAL: NCT06138912
Title: Normal Functional Local Alignment and Segmental Motion at the Thoracolumbar Junction: A Cross-Sectional Study of Healthy Subjects
Brief Title: Thoracolumbar Junction
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Han Moon-Soo, Department of Neurosurgery, Chonnam National University Hospital
Other Study IDs: ChonnamNUH
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Spinal Curvatures
Keywords: Thoracolumbar spine; Alignment; Range of motion
MeSH Terms: conditions — Spinal Curvatures | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Age: 20-29, 30-39, 40-49, 50-59, 60-69, and 70-79
  Interventions: Radiation: plain radiography (x-ray)
- sex: each group included 10 subjects
  Interventions: Radiation: plain radiography (x-ray)

INTERVENTIONS:
Radiation: plain radiography (x-ray) — Radiographic imaging of the subjects was performed, and anteroposterior, lateral, flexion-extension, and right-left lateral bending radiograph views were obtained

SUMMARY:
Several studies have investigated the mechanical behavior of the thoracolumbar spine. However, an accurate reference for normal functional local alignment and segmental motion at the thoracolumbar junction is still illusive. Therefore, we conducted a cross-sectional cohort study with a balanced distribution of age and sex of healthy subjects to examine the normal alignment and segmental motion at the thoracolumbar junction using dynamic plain radiography. This study aimed to provide data that can be used when planning surgery or performing rehabilitation in pathological situations.

ELIGIBILITY:
Inclusion Criteria:

* A total of 120 asymptomatic healthy volunteer subjects aged 20 to 79 without back pain complaints were included if they successfully met the study's exclusion criteria

Exclusion Criteria:

* (1) coronal deformity (Cobb angle > 10°); (2) a history of prior spine surgery; (3) a history of hip or knee arthroplasty or any other realignment surgery of the lower extremities (osteotomy, trauma, etc.); (4) complaints of back or neck pain that resulted in missed work, affected daily living activities, participation in recreational activities or required narcotic pain medication; (5) degenerative or pathologic conditions of the spine that necessitated physician intervention (i.e., physician appointment or epidural steroid injections); (6) non-ambulatory patients; (7) a history of neuromuscular disorders, inflammatory arthritis, or congenital anomalies; and (8) pregnancy

Ages: 20 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 120 asymptomatic healthy volunteer subjects aged 20 to 79 without back pain complaints
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Normal Functional Local Alignment and Segmental Motion at the Thoracolumbar Junction | 2year
  The present study measured the normal functional Local Alignment and Segmental Motion at the Thoracolumbar junction based on the age and sex of healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hospital, Gwangju, Dong-gu, South Korea

IPD SHARING:
Plan to Share IPD: No